CLINICAL TRIAL: NCT07073989
Title: Investigating the Impact of Afferent Stimulation on Proprioceptive Function in Post-Stroke Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Julio S. Lora Millán (Other)
Responsible Party: Sponsor-Investigator, Julio S. Lora Millán, Principal Investigator, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeuroBot_ESNA_v1
Record Dates: First submitted 2025-06-20; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Healthy Subjects or Volunteers; Chronic Stroke
Keywords: Afferent stimulation; Proprioception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects (Experimental): Intervention applied to healthy subjects
  Interventions: Device: Afferent stimulation
- Stroke patients (Experimental): Stimulation applied to stroke patients
  Interventions: Device: Afferent stimulation

INTERVENTIONS:
Device: Afferent stimulation — Stimulation applied through mechanical vibration or low-intensity electric currents

SUMMARY:
The objective of this study is to assess the functionality of a sensory stimulation device that uses mechanical vibrations and low-intensity electrical currents to deliver proprioceptive feedback to stroke patients regarding their movements.

ELIGIBILITY:
Inclusion Criteria:

* For healthy subjects:

  1. No neurological or orthopedic conditions affecting upper limb movement.
  2. No surgical interventions on the upper limbs within the past 6 months.
  3. General physical condition adequate to perform the session.
  4. Cognitive abilities sufficient to understand and carry out the experimental procedure.
* For stroke survivors:

  1. Ischemic or hemorrhagic stroke resulting in motor impairments in the upper limb.
  2. Chronic stroke condition.
  3. Subjects with sufficient cognitive abilities to follow instructions and actively participate in the therapy.
  4. Mini-Mental State Examination (MMSE) score > 24.
  5. Subjects presenting hemiparesis and mild-to-moderate impairment in the upper limb (score on the Fugl-Meyer Motor Assessment for the upper limb, sections A-D, between 35 and 53 points). The maximum score on the FM scale is 66, with the following severity classifications:
* 0-15: severe impairment
* 16-34: moderate-to-severe impairment
* 35-53: mild-to-moderate impairment
* 54-66: mild impairment 6. Subjects presenting upper limb hypertonia with a score below 3 on the Modified Ashworth Scale.

  7. Subjects who have signed the informed consent document to voluntarily participate in the experiments.

Exclusion Criteria:

1. Acute musculoskeletal disorders.
2. Peripheral vascular diseases.
3. Acute cardiopulmonary conditions.
4. Acute neurological disorders.
5. Restricted mobility of upper limb joints due to any cause.
6. Pain as a cause of impaired upper limb mobility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Motor illusion | Periprocedural
  Motor illusion is evaluated by instructing the patient to replicate the movement they experienced in the contralateral limb. Inertial sensors will be placed in such limb to acquire the movement performed by the subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Móstoles, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided